CLINICAL TRIAL: NCT06432400
Title: Identification of Post-Traumatic Stress Disorder in Adult Patients With Substance Use Disorders Followed up in the Medical and Psychological Centre: Multicentre Descriptive Study
Brief Title: Identification of Post-Traumatic Stress Disorder in Adult Patients With Substance Use Disorders
Acronym: IRTIPAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Refusal by the Ethics Committee
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRD0824; 2024-A00790-47 (Other: ANSM)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-05

CONDITIONS: Trauma
Keywords: Post Traumatic Stress Disorder; Complex post traumatic stress disorder; Medical and Psychological Centre
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Substance use disorders (Other): Group composed of patients suffering from disorders related to the use of alcohol, cannabis, opiates, inhalants, sedatives, hypnotics, anxiolytics, stimulants, hallucinogens (all of these disorders will have been diagnosed by a doctor before or during follow-up according to Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM 5) criteria)
  Interventions: Other: Patient questionnaires

INTERVENTIONS:
Other: Patient questionnaires — Patients questionnaires, on paper and data collection on patients medical file

SUMMARY:
The aim of this study is to show that early identification of PTSD and CPTSD would increase recognition of these disorders and facilitate diagnosis, referral and recovery.

DETAILED DESCRIPTION:
Between 61% and 81% of men and 51% to 74% of women are exposed to a traumatic event in their lifetime. These events may be brief and discrete, prolonged and/or recurrent, and may be direct or indirect. Direct or indirect exposure to traumatic events can lead to serious negative psychological consequences, including post-traumatic stress disorder (PTSD) and complex post-traumatic stress disorder (CPTSD). People exposed to complex traumatic events are at risk not only of suffering from PTSD or Complex PTSD, but also from other mental health co-morbidities, such as substance use disorders (drugs, alcohol, benzodiazepine misuse) , often associated with the repetition of situations of interpersonal violence from which it is difficult, if not impossible, to escape.

Caring for people suffering from psychological trauma is a major public health issue. However, there are no good clinical practice guidelines for diagnosis, assessment and treatment, which would enable good practice to be standardised and disseminated. The prevention, detection, early support and appropriate guidance of people suffering from post-traumatic sequelae promote their recovery and improve their quality of life. The World Health Organization (WHO) refers to this as psychological distress, and points out that if it is not properly identified or accompanied, it can tip a person into illness or increase social difficulties. When it is temporary and follows a stressful event, it is considered a normal adaptive reaction. On the other hand, when it becomes intense and persistent, it may be an indicator of a psychological disorder. The public health challenge associated with PTSD is to better recognise, diagnose and treat it, as it can have serious consequences for the quality of life, social functioning and suicide risk of those affected.

The aim of this study is to show that early identification of PTSD and CPTSD would increase recognition of these disorders and facilitate diagnosis, referral and recovery. It would also make it possible to provide individualised support for patients and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria :

* Patient aged 18 or over
* Patient followed up at the adult Medical and Psychological Centre in the centres taking part in the study
* Patient suffering from disorders related to the use of alcohol, cannabis, opiates, inhalants, sedatives, hypnotics, anxiolytics, stimulants, hallucinogens (all of these disorders will have been diagnosed by a doctor before or during follow-up according to DSM 5 criteria).
* Patient aware of their substance use disorders
* Patient informed and did not object to participating in the study

Exclusion Criteria :

* Patient previously diagnosed with PTSD or CPTSD
* Patient agitated and/or aggressive
* Patient under guardianship/curators
* Patient who do not speak or understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the proportion of Post-Traumatic Stress Disorder (PTSD) in patients with substance use disorders | At the end of the study, an average of 12 month
  Percentage of patients with PTSD among those with substance use disorders Patients with PTSD will be identified using the International Trauma Questionnaire (ITQ) : A diagnosis of PTSD requires the presence of at least one symptom in each of the following dimensions
  * P1 or P2 ≥ 2
  * P3 or P4 ≥ 2
  * 5 or P6 ≥ 2 AND
  * P7 or P8 or P9 ≥ 2
  Score ITQ for PTSD : ≥ 8

SECONDARY OUTCOMES:
Distinguishing between the prevalence of Post-Traumatic Stress Disorder (PTSD) and Complex Post-Traumatic Stress Disorder (CPTSD) | At the end of the study, an average of 12 month
  Percentage of patients with CPTSD among those with substance use disorders Patients with CPTSD will be identified using the International Trauma Questionnaire (ITQ) : A diagnosis of CPTSD requires a PTSD : ≥ 8 and, at least, one symptom in each of the dimensions of disturbance of self-organisation
  * C1 or C2 ≥ 2
  * C3 or C4 ≥ 2
  * C5 or C6 ≥ 2 AND
  * C7 or C8 or C9 ≥ 2
  Score ITQ for CPTSD : ≥ 16
Identification of risk factors by comparing demographic data of PTSD versus CPTSD patients | At the end of the study, an average of 12 month
  Risk factors will be identified from the demographic data collected via the patient characteristics questionnaire between PTSD and CPTSD patients
Identification of the pathologies most associated with PTSD and CPTSD | At the end of the study, an average of 12 month
  The pathologies most frequently associated with PTSD and CPTSD will be identified by collecting the pathologies present in the medical records of all patients.
Comparison of the time between management and identification of patients with PTSD versus CPTSD | At the end of the study, an average of 12 month
  Comparison for number of days between the start of treatment for substance use disorders and the identification of PTSD or CPTSD

CONTACTS AND LOCATIONS:
Overall Officials: Déborah DELABY, Principal Investigator — Isarien Hospital Centre
Locations (2):
- France (2):
  - Medical and Psychological Centre - Novo Hospital - Site Beaumont-sur-Oise, Beaumont-sur-Oise
  - Medical and Psychological Centre - Isarien Hospital Centre, Clermont